CLINICAL TRIAL: NCT07135726
Title: OpenNOTES: Online Access to Clinical Treatment Notes for Outpatients - an Interventional, Prospective, Controlled Mixed-methods Study
Brief Title: Online Access to Clinical Treatment Notes for Outpatients
Acronym: OpenNOTES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julian Schwarz (Other)
Collaborators: Universität zu Köln (Unknown); Technische Hochschule Brandenburg (Unknown)
Responsible Party: Sponsor-Investigator, Julian Schwarz, Julian Schwarz, MD Specialist in Psychiatry and Psychotherapy, Research Associate Mental Health Policy & Digitization Research Group, Medizinische Hochschule Brandenburg Theodor Fontane
Organization: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 271012025-BO-E
Record Dates: First submitted 2025-06-16; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Mental Disorders; Chronic Disease; Primary Health Care; Outpatients; Internal Medicine; Aged; Comorbidity
MeSH Terms: conditions — Mental Disorders; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Notes Access (Experimental)
  Interventions: Device: Patient Portal-Based Access to Clinical Notes
- No Notes Access (No Intervention): Due to potential selection bias of the intervention group, which occurs due to voluntary participation in the intervention, a control group is surveyed at t0, which does not participate in the intervention, so that an adjustment for the systematic differences, if any, between the intervention and control group is possible at t0. The survey of a post-intervention control group (t1) serves to adjust for any time-varying effects so that a general time effect can be ruled out.
  n=91 patients with a pre-intervention and a post-intervention control group of n=91 patients

INTERVENTIONS:
Device: Patient Portal-Based Access to Clinical Notes — An intra-individual comparison of patient-reported outcomes is planned for the intervention group. For this purpose, the pre-intervention survey of the intervention group is conducted upon inclusion in the study, the post-intervention survey at the earliest after the intervention has been used once (accessing their open note). Due to potential selection bias of the intervention group, which occurs due to voluntary participation in the intervention, a control group is surveyed at t0, which does not participate in the intervention, so that an adjustment for the systematic differences, if any, between the intervention and control group is possible at t0. The survey of a post-intervention control group (t1) serves to adjust for any time-varying effects so that a general time effect can be ruled out.
  Arms: Shared Notes Access

SUMMARY:
This study investigates the feasibility and impact of patient access to clinical notes written by their healthcare providers-a concept known as Open Notes. While international research has already demonstrated positive effects of Open Notes on patient empowerment and treatment outcomes, there is a lack of corresponding evidence for the German healthcare context. The quasi-experimental study therefore combines quantitative and qualitative methods to evaluate the effects of Open Notes on patient-reported outcomes as well as clinical practice.

The study is structured into five modules, each addressing specific research questions:

Module A - Summative Outcome Evaluation in Patients: Does the use of Open Notes lead to a significant increase in patient-reported outcomes such as empowerment and self-efficacy? Module B - Formative Process Evaluation with Stakeholders: What experiences do patients, relatives and clinicians have with Open Notes and what challenges and barriers arise in their use? Module C - Changes in Clinical Documentation: How do language style and content of clinical notes change when they are shared with patients as Open Notes? Module D - Optimization through Artificial Intelligence: Can clinical notes be processed using artificial intelligence in a way that makes them easier for patients to understand compared to conventional medical documentation? Module E - Integration into National Data Infrastructure: What technical, organizational and legal requirements must be met to successfully integrate Open Notes into the national telematics infrastructure and the electronic health record or routine care? The overall goal is to identify both patient-related outcomes and structural conditions for the sustainable implementation of Open Notes in the German healthcare system. The use of artificial intelligence is intended to further enhance patient-centeredness while reducing the burden on clinical staff.

ELIGIBILITY:
Inclusion Criteria:

Patients (General, Module A & D):

* Aged 18 years or older
* Outpatient treatment at one of the four study centers
* For intervention group: access to an internet-enabled device (e.g. smartphone, tablet, computer) and ability to receive text messages

For Module D:

* Experience with the respective disease or medical field (e.g. via prior treatment experience or basic medical understanding)
* At least one documented clinical treatment in the internal system of a participating center within the 12 months prior to intervention start
* Availability of clinically relevant treatment notes (e.g. physician letters, progress notes, discharge summaries, consultation notes) suitable for anonymized analysis

Patients (Control Group - Module A):

•No requirement for access to an internet-enabled device

Healthcare Practitioners (Modules A & D):

* Aged 18 years or older
* Employed at one of the study centers
* Ability to give informed consent
* For Module D: experience in relevant clinical field and familiarity with medical terminology and treatment standards

Relatives (Module B):

* Aged 18 years or older
* Ability to give informed consent
* Identified as family member, friend, or legal representative of a participating patient

Experts (Module E):

* Demonstrated expertise or professional experience in digital health Relevant experience with telematics infrastructure (TI), HL7 FHIR®, ePA, KIM, TIM, or affiliation with relevant institutions (e.g. gematik GmbH, HL7 Deutschland e.V., mio42 GmbH)
* Participation in or co-design of health IT interoperability projects

Patients and Physicians (Module E):

* Good proficiency in German (workshops conducted in German)
* Basic digital literacy and experience with digital technologies in healthcare

Exclusion Criteria:

General:

* Insufficient German language skills
* Severe organic brain disorders with cognitive impairment
* Intellectual disability
* Acute self-endangerment or danger to others at time of inclusion
* Lack of capacity to provide informed consent
* Lack of access to an internet-enabled device and inability to receive text messages (except in control group of Module A)

Module D:

* Clinical notes that cannot be anonymized due to legal, ethical, or technical restrictions
* Presence of rare diagnoses or unique treatment histories that hinder effective anonymization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1092 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Empowerment Measured by the Health Care Empowerment Inventory | From baseline to follow-up, up to 24 months per participant in the intervention group
  This primary outcome measures change in patient empowerment using the Health Care Empowerment Inventory. The HCEI is a validated self-report instrument assessing a patient's sense of being informed, engaged, committed, collaborative, and tolerant of uncertainty in relation to their health care. Scores range from 1 to 5 per item and are aggregated for a total score. Data will be collected via the PEPPPSY patient portal before and after the first access to Open Notes. Analyses include intra-individual pre/post comparisons in the intervention group and comparisons with a non-exposed control group. Outcome modeling will take frequency of Open Notes use into account.
Stakeholder Experiences with Open Notes Assessed by Semi-Structured Interviews and Focus Groups Using a CFIR-Based Guide | Four iterative sampling points over a 20-month period (t0 to t3, in 3-month intervals)
  This outcome captures user experiences with Open Notes, including knowledge and beliefs about the intervention, attitudes toward digital access to clinical notes, and digital literacy. Data will be collected through 88 semi-structured interviews (44 patients, 20 relatives, 24 practitioners) and 16 focus groups (~80 participants), guided by an interview protocol based on the Consolidated Framework for Implementation Research (CFIR). This topic is primarily addressed in the interviews. Data will be analyzed using qualitative content analysis.
Perceived Advantages and Challenges of Open Notes Assessed by Semi-Structured Interviews and Focus Groups Using a CFIR-Based Guide | Four iterative sampling points over a 20-month period (t0 to t3, in 3-month intervals)
  This outcome explores stakeholder views on the benefits and challenges of using Open Notes. Topics include perceived usefulness, empowerment, relative advantages, usability, and individual characteristics such as health literacy. Data will be collected through 88 semi-structured interviews and 16 focus groups using a CFIR-based guide. This outcome is primarily addressed in the interviews. Data will be analyzed using qualitative content analysis.
Impact of Open Notes on Therapeutic Relationship and Communication Assessed by Semi-Structured Interviews and Focus Groups Using a CFIR-Based Guide | Four iterative sampling points over a 20-month period (t0 to t3, in 3-month intervals)
  This outcome investigates how stakeholders perceive changes in therapeutic relationships and communication following the introduction of Open Notes. Topics include mutual trust, shared decision-making, and the involvement of relatives. Data are collected through semi-structured interviews and focus groups using a CFIR-based guide. This topic is primarily addressed in the interviews. Data will be analyzed using qualitative content analysis.
Perspectives on Future Implementation of Open Notes Assessed by Semi-Structured Interviews and Focus Groups Using a CFIR-Based Guide | Four iterative sampling points over a 20-month period (t0 to t3, in 3-month intervals)
  This outcome captures stakeholder perspectives on the future integration of Open Notes into routine care. Topics include attitudes toward adoption, digital competencies, organizational readiness, infrastructure requirements, and implementation support needs (e.g., training, design adjustments). Data will be collected via semi-structured interviews and 16 focus groups using a CFIR-based guide. This outcome is primarily addressed in the focus groups. Data will be analyzed using qualitative content analysis.
Change in Linguistic Complexity of Clinical Notes Measured by Flesch-Kincaid Readability Index | 6 months for pre-Open Notes documentation and 6 months for post-Open Notes documentation
  This outcome assesses changes in linguistic complexity of clinical notes before and after Open Notes implementation using the Flesch-Kincaid readability index. A total of 20 notes before and 20 after implementation will be analyzed per study center using an online tool (https://conrics.com/features/). Higher scores indicate easier readability. Results will be compared across timepoints and study sites.
Change in Length of Clinical Notes Measured by Word and Sentence Count | 6 months for pre-Open Notes documentation and 6 months for post-Open Notes documentation
  This outcome examines changes in the average length of clinical notes before and after Open Notes implementation. Word and sentence counts will be determined for 20 notes before and 20 after implementation per study center. Descriptive and inferential comparisons will be made between groups.
Change in Thematic Content of Clinical Notes Measured by Linguistic Inquiry and Word Count (LIWC) | 6 months for pre-Open Notes documentation and 6 months for post-Open Notes documentation
  This outcome investigates whether the thematic focus of clinical notes changes following the implementation of Open Notes. LIWC software will be used to analyze 20 notes before and 20 after implementation per study center. Changes in thematic categories such as affective tone, cognitive processing, and personal pronouns will be examined and compared descriptively.
Readability of AI-Modified vs. Original Clinical Notes Rated by Patients Description | 27 months (including chatbot testing, AI modification of notes, and data collection)
  This outcome assesses whether AI-modified clinical notes are rated as more readable than original notes. A total of 400 anonymized notes from the 12 months before the Open Notes rollout will be processed using large language models (e.g., ChatGPT, Neuroflash). Readability will be evaluated by patients using the Patient Education Materials Assessment Tool (PEMAT) and the Flesch-Kincaid Grade Level.
Perceived Information Quality of AI-Modified vs. Original Clinical Notes Rated by Patients Description | 27 months (including chatbot testing, AI modification of notes, and data collection)
  This outcome assesses whether AI-modified clinical notes are rated as providing higher-quality information compared to original notes. A total of 400 anonymized notes from the 12 months before the Open Notes rollout will be processed using large language models (e.g., ChatGPT, Neuroflash). Perceived information quality will be measured by patients using selected items from the Health Information National Trends Survey (HINTS).
Subjective Understanding of AI-Modified vs. Original Clinical Notes Rated by Patients Description | 27 months (including chatbot testing, AI modification of notes, and data collection)
  This outcome assesses whether AI-modified clinical notes are rated as more understandable than original notes. A total of 400 anonymized notes from the 12 months before the Open Notes rollout will be processed using large language models (e.g., ChatGPT, Neuroflash). Subjective understanding will be evaluated by patients using the Single Item Literacy Screener (SILS) and brief comprehension tasks.
Technical and Organizational Requirements for Integrating Open Notes into the German Telematics Infrastructure (TI) and Electronic Health Record (ePA) | Up to 23 months
  This module will produce technical and legal specifications for integrating Open Notes into the German national telematics infrastructure (TI), including the electronic patient record (ePA), the KIM communication system, and the TIM messaging service. Integration prototypes will be developed in three design thinking workshops (6-8 experts and 4 users each), ensuring HL7 FHIR® compliance. A Delphi-like process will generate and rate implementation concepts. Measured outcomes will include the number and type of integration use cases, HL7 FHIR® conformance levels, and expert consensus scores for each proposed concept. All results will align with existing interoperability and legal standards.

SECONDARY OUTCOMES:
Change in Shared Decision Making Measured by the 9-Item Shared Decision Making Questionnaire (SDM-Q-9) | From baseline to follow-up, up to 24 months per participant in the intervention group
  Assesses perceived shared decision making using the SDM-Q-9. This 9-item self-report instrument uses a 6-point Likert scale and is transformed to a 0-100 total score, with higher scores indicating more shared decision making. Data will be collected via the PEPPPSY patient portal before and after first access to Open Notes. Analyses include intra-individual pre/post comparisons and comparisons with a non-exposed control group. Outcome modeling will take frequency of use into account.
Change in Self-Efficacy Measured by the General Self-Efficacy Scale (GSE) | From baseline to follow-up, up to 24 months per participant in the intervention group
  Assesses perceived self-efficacy using the General Self-Efficacy Scale, a 10-item measure scored from 1 to 4. Total scores range from 10 to 40, with higher scores indicating stronger self-efficacy expectations. Data will be collected via the PEPPPSY portal before and after first access to Open Notes. Analyses include intra-individual and between-group comparisons. Outcome modeling will account for usage frequency.
Change in Perceived Disease Management Measured by the EFK-HPC (Effektivität der Krankheitsbewältigung - Hochproblematische Chronizität) | From baseline to follow-up, up to 24 months per participant in the intervention group
  Assesses coping strategies in patients with chronic illness using the EFK-HPC scale, a validated instrument designed to measure the effectiveness of coping with difficult chronic conditions. Items are rated on Likert scales; higher scores reflect better disease management. Data will be collected via the PEPPPSY portal pre- and post-intervention. Analyses include intra-individual and between-group comparisons; outcome modeling includes usage frequency.
Change in Patient Satisfaction Measured by the ZUF-8 Questionnaire | From baseline to follow-up, up to 24 months per participant in the intervention group
  Assesses patient satisfaction using the ZUF-8, a validated short version of the Client Satisfaction Questionnaire (CSQ-8), with 8 items rated on a 4-point scale. Higher total scores indicate greater satisfaction with care. Data will be collected via the PEPPPSY portal before and after access to Open Notes. Analyses include intra-individual comparisons and group-level modeling that incorporates usage frequency.
Clarity, Accuracy, and Appropriateness of AI-Modified vs. Original Clinical Notes Rated by Health Professionals | 27 months (including chatbot testing, AI modification of notes, and data collection)
  This outcome assesses whether AI-modified clinical notes are rated as clearer, more accurate, and more appropriate than original notes. A total of 400 anonymized notes from the 12 months before the Open Notes rollout will be processed using large language models (e.g., ChatGPT, Neuroflash). Health care professionals will evaluate the notes using a modified DISCERN Instrument and structured evaluation forms.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Wurster, M.Sc. Health Services Research, Study Director — University of Cologne; Eva Meier-Diedrich, M.Sc. Psychology, Study Director — Medical School Brandenburg; Julian Schwarz, MD, Specialist in Psychiatry, Principal Investigator — Medical School Brandenburg; Ute Karbach, Priv.-Doz. Dr. rer. pol., Principal Investigator — University of Cologne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Johnson MO, Rose CD, Dilworth SE, Neilands TB. Advances in the conceptualization and measurement of Health Care Empowerment: development and validation of the Health Care Empowerment inventory. PLoS One. 2012;7(9):e45692. doi: 10.1371/journal.pone.0045692. Epub 2012 Sep 19. PMID 23029184
- [Background] Wurster, Florian, Eva Meier-Diedrich, I. Demirer, Catherine DesRoches, Nina Goldberg, Maria Hägglund, C. Herrmann, U. Karbach, A. Purohit, T. Schrader, J. Schwarz, 2024. "Online-Zugang Zu Klinischen Behandlungsnotizen Für Ambulant Versorgte Patienten (Studienprotokoll Zur OpenNOTES-Studie)." Nervenheilkunde, 43(12), 714-719.
- See also: General information about the concept of open notes itself and the OpenNOTES-study — https://www.opennotes.info/en/